CLINICAL TRIAL: NCT00736372
Title: A Phase Ib Trial of PX-12 Administered as a 72-Hour Infusion Every 21 Days in Patients With a Histologically or Cytologically Confirmed Diagnosis of Advanced or Metastatic Cancer That is Refractory to Standard Treatment
Brief Title: A Trial of PX-12 in Patients With a Histologically or Cytologically Confirmed Diagnosis of Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cascadian Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PX-12-004
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2013-03

CONDITIONS: Metastatic Cancer; Advanced Cancer
Keywords: cancer; metastatic cancer; advanced or metastatic cancer
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigational Drug (Experimental): Dose Escalation
  Interventions: Drug: PX-12

INTERVENTIONS:
Drug: PX-12 — Intravenous infusion, dose escalation, infused over a 72 hour period on days 1, 2 and 3 of a 21-day cycle until progression or development of unacceptable toxicity

SUMMARY:
PX-12 (1-methylpropyl 2-imidazolyl disulfide) is a novel small molecule inhibitor of thioredoxin-1, a small protein over-expressed in many human cancers that is associated with aggressive tumor proliferation, angiogenesis, and drug resistance. This study is being conducted to determine the maximally tolerated dose of PX-12 delivered as a 72-hour infusion over days 1, 2, and 3 of a 21-day cycle in patients with advanced or metastatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed diagnosis of advanced or metastatic cancer or lymphoma whose tumors are refractory to standard therapy or for whom no standard therapy is available that increases survival by at least three months.
2. Men and women at least 18 years of age.
3. A predicted life expectancy of at least 12 weeks.
4. ECOG performance status of 0-2 .
5. Patients must have discontinued previous anticancer therapy and/or other investigational agents at least three weeks prior to treatment with PX-12 (six weeks for mitomycin C and nitrosureas) and recovered (grade 1 or less) from the toxic effects of that treatment. In the case of oral agents with a short half life, on a case by case basis, a minimum of a two week interval may be permitted.
6. Patients must have discontinued any radiation therapy at least four weeks prior to treatment with PX-12 and have recovered from all radiation-related toxicities. Palliative radiation of 10 fractions or less is permitted and a four week interval is not necessary (also allowed during therapy).
7. The patient has adequate hematologic function as defined by the following:

   platelets >100,000/μL; hemoglobin >9 g/dL (may be transfused to this level); ANC > 1,500 cells/μL.
8. The patient has adequate hepatic function as defined by the following: bilirubin <2.0 mg/dL;aspartate aminotransaminase (AST/SGOT) & alanine aminotransferase (ALT/SGPT) <2.5 times (or up to five ULN for patients with liver metastases) institutional upper limit of normal (ULN). International Normalized Ratio (INR) and activated partial thromboplastin time (aPTT) within 1.5 times ULN unless subject is on coumadin.
9. The patient has adequate renal function as defined by serum creatinine level

   ≤ 1.5 x ULN.
10. Patient has signed informed consent.
11. Patient is compliant with the study and in geographic proximity to allow adequate follow-up.
12. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method; abstinence) prior to study entry and for the duration of study participation. Childbearing potential will be defined as women who have had menses within the past 12 months, who have not had tubal ligation or bilateral oophorectomy. Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician

Exclusion Criteria:

1. Patients with symptomatic pulmonary disease, e.g., active chronic obstructive/restrictive pulmonary disease, asthma, evidence of interstitial pneumonitis, pulmonary fibrosis, etc.
2. Patients with history of dyspnea, dyspnea on exertion, or paroxysmal nocturnal dyspnea.
3. Patients that meet the Medicare criteria for receiving home oxygen or are on oxygen.
4. Patients with a history of prior lung radiation.
5. Patients with any active infection requiring i.v. antibiotics at study entry.
6. Any serious concomitant systemic disorders that in the opinion of the investigator would place the patient at excessive or unacceptable risk of toxicity.
7. Significant central nervous system or psychiatric disorder(s) that preclude the ability of the patient to provide informed consent.
8. Known or suspected brain metastases that have not received adequate therapy. In the case of previously treated brain metastases, a minimum of four weeks interval between completion of radiation therapy and registration on study with radiologic evidence of stable or responding brain metastases is required. In the setting of previous CNS metastasectomy, adequate (minimum four week) recovery from surgery and/or radiation therapy should be documented.
9. Major surgery within four weeks of treatment with PX-12.
10. Patients with a history of seizures.
11. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
12. Patients who are breastfeeding or pregnant (confirmed by serum β-HCG within 10 days prior to the start of study treatment if applicable).
13. Any condition that could jeopardize the safety of the patient and compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To determine the MTD of PX-12 delivered as a 72-hour infusion over days 1, 2, and 3 of a 21-day cycle | 21 days

SECONDARY OUTCOMES:
When delivered as a 72 hour intravenous infusion on days 1, 2, and 3 of a 21-day cycle: Evaluate the safety profile of PX-12 | 42 days
When delivered as a 72 hour intravenous infusion on days 1, 2, and 3 of a 21-day cycle: Assess the pharmacodynamics of PX-12 using surrogate tissues obtained pre- and post-drug treatment | 42 days
When delivered as a 72 hour intravenous infusion on days 1, 2, and 3 of a 21-day cycle: Assess pharmacokinetic profiles of PX-12 in plasma samples | 42 days
When delivered as a 72 hour intravenous infusion on days 1, 2, and 3 of a 21-day cycle: Identify any antitumor activity of PX-12 in this patient population | 42 days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - TGen Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Tyler Cancer Center, Tyler, Texas